CLINICAL TRIAL: NCT06604949
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Dose of LP-003 in Healthy Adult Subjects
Brief Title: A Study of Single Dose of LP-003 in Healthy Adult Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10-LP003-07
Record Dates: First submitted 2024-09-14; First posted 2024-09-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP-003 (Experimental): Single dose administration, with a dosage of 200 mg LP-003
  Interventions: Drug: LP-003 200mg
- Placebo (Placebo Comparator): Single dose administration of LP-003 placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LP-003 200mg — Subcutaneous injection of 200 mg LP-003
  Arms: LP-003
Drug: Placebo — Subcutaneous injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of LP-003 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged ≥18 and ≤ 50 years.
2. Male subjects must weigh ≥50 kg, and female subjects must weigh ≥45 kg, with a BMI between 19.0 and 28.0 kg/m² (inclusive).
3. Male subjects and their partners or female subjects must agree to use one or more non-pharmaceutical contraceptive methods (such as total abstinence, condoms, Iuds, partner ligation, etc.) during the trial period and for 6 months after the trial, and do not plan to donate sperm or eggs.
4. The subjects fully understand the purpose, nature, method and possible adverse reactions of the experiment, and voluntarily participate in the experiment and sign the informed consent.
5. The subjects were able to communicate well with the researchers and complete the study according to the protocol.

Exclusion Criteria:

1. People who are allergic to the experimental drug and any of its excipients, have a history of allergy to monoclonal antibodies, and are allergic to multiple drugs and food.
2. Patients who have been or are currently suffering from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatric and metabolic abnormalities, or any other diseases that can interfere with the test results.
3. Patients who had undergone surgery within 3 months before the trial that the researchers judged would affect drug absorption, distribution, metabolism, and excretion, or had surgery within 4 weeks prior to the trial, or planned to have surgery during the study period.
4. Any history of infection within 14 days prior to administration.
5. A person who is currently infected with parasites or has traveled to an endemic area within the last 3 months or 24 weeks prior to administration.
6. Pregnant and lactating women.
7. Hepatitis B surface antigen, hepatitis C virus antibodies, human immunodeficiency virus antibodies, treponema pallidum antibodies A positive person.
8. Patients who have received any biological agent (including antibodies or derivatives such as omazumab) within 16 weeks prior to administration (or 5 half-lives, selecting the longer time period).
9. Participants who had participated in other clinical trials within 3 months prior to screening.
10. The investigator deems any condition unsuitable for study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | From the beginning of first patient in (FPI) to the end of study up to approximately 12 months

SECONDARY OUTCOMES:
Area under the concentration-time curve from the first dose to the last measurable concentration time (AUC0-t) | From the beginning of first patient in (FPI) to the end of study up to approximately 12 months
The proportion of ADA (Anti Drug Antibody) positive subjects | From the beginning of first patient in (FPI) to the end of study up to approximately 12 months
Serum total IgE and free IgE levels compared to baseline | From the beginning of first patient in (FPI) to the end of study up to approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No